CLINICAL TRIAL: NCT06761677
Title: A Multi-Center, Global, Open-Label, Phase 1b/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Intravenous Brincidofovir in Patients With Relapsed or Refractory Lymphoma As Well As to Evaluate the Safety and Efficacy of Intravenous Brincidofovir in Patients With Relapsed or Refractory Extranodal Natural Killer/T-cell Lymphoma Using The Recommended Phase 2 Dose
Brief Title: A Phase 1b/2 Study of Intravenous Brincidofovir in Patients With Relapsed or Refractory Lymphoma and Relapsed or Refractory Extranodal Natural Killer/T-cell Lymphoma
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to challenges in recruiting eligible patients under the protocol.
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCV-NL01
Record Dates: First submitted 2024-12-24; First posted 2025-01-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Lymphoma Including ENKL
Keywords: SyB V-1901; BCV; Relapsed or refractory Lymphoma; Extranodal Natural Killer/T-cell Lymphoma; ENKL; EBV-positive nodal T- and NK-cell lymphoma; EBV + nTNKCL; nodal T-follicular helper cell lymphoma; nTFHcL; angioimmunoblastic T-cell lymphoma; AITL; peripheral T-cell lymphoma not otherwise specified; PTCL-NOS; anaplastic large cell lymphoma; ALCL; diffuse large B-cell lymphoma; DLBC; DLBCL-NOS; adult T-Cell Leukemia Lymphoma; ATLL
MeSH Terms: conditions — Recurrence; Lymphoma; Epstein-Barr Virus Infections; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia-Lymphoma, Adult T-Cell | interventions — brincidofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brincidofovir twice weekly (BIW) via intravenous infusion (Experimental)
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — Phase 1b part is dose escalation study evaluating three dose levels of BCV, and participants will be assigned to a dose schedule in the order of study entry. In Phase 2 part, participants will receive BCV BIW at the RP2D (determined in the Phase 1b part).
  Other Names: SyB V-1901; BCV

SUMMARY:
This study is a multi-center, global, open-label, Phase 1b/2 clinical study, and it will be conducted at multiple study sites in several countries, including Japan, Korea, and Singapore, to reveal the safety, tolerability, dose limiting toxicity (DLT), maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D), pharmacokinetics (PK), and preliminary efficacy of BCV in patients with relapsed or refractory lymphoma and to assess the efficacy and safety of Brincidofovir (SyB V-1901, BCV) in patients with relapsed or refractory Extranodal Natural Killer/T-cell Lymphoma (ENKL).

This study consists of 2 parts and will enroll a total (maximum) of 43 male and female participants who meet the eligibility criteria (Phase 1b part: Up to 18 participants [3 to 6 participants in each of the 3 cohorts], Phase 2 part: 25 participants).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are histopathologically diagnosed with ENKL based on the World Health Organization (WHO) Classification of Malignant Lymphoma 5th Edition (WHO-HAEM5) (can be enrolled in the Phase 1b part and the Phase 2 part) or patients diagnosed with EBV-positive nodal T- and NK-cell lymphoma (EBV + nTNKCL), nodal T-follicular helper cell lymphoma (nTFHcL) (including angioimmunoblastic T-cell lymphoma (AITL) as defined in the WHO Classification, 4th Edition), peripheral T-cell lymphoma not otherwise specified (PTCL, NOS), anaplastic large cell lymphoma (ALCL), diffuse large B-cell lymphoma (DLBCL) (e.g., DLBCL, NOS), or adult T-Cell Leukemia Lymphoma (ATLL) (can only be enrolled in the Phase 1b part)
* Patients with relapsed or refractory lymphoma and previously treated with systemic chemotherapy (history of multidrug chemotherapy including L-asparaginase such as SMILE therapy for ENKL is mandatory) who are ineligible for other systemic therapies
* Patients with the following Eastern Cooperative Oncology Group (ECOG) Performance Status (PS):
* Phase 1b part: 0-1
* Phase 2 part: 0-2

Exclusion Criteria:

* Patients with another active malignant tumor requiring treatment
* Patients with NCI-CTCAE Grade 2 or higher diarrhea (increase of 4 or more bowel movements per day compared to usual number of bowel movements) within 7 days prior to starting the first dose of BCV
* Graft-Versus-Host Disease (GVHD) patients requiring immunosuppressive agents
* Patients with a history of Cidofovir intolerance
* Patients with a history of being diagnosed with cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-10-23 (Estimated); Study Completion 2029-05-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1b part (Dose Escalation Part) | 28 days
  Adverse events (AEs) that meet the protocol-defined DLT criteria in Cycle 1 and the number of participants that developed these AEs
Phase 2 part (Expansion Part) | 7 months
  Best Overall Response as of end of treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Queen Mary Hospital, Hong Kong, China
- Japan (6):
  - Tokyo Metropolitan Komagome Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūōku
  - Cancer Institute Hospital Of JFCR, Kōtoku
  - Kyoto University Hospital, Kyoto
  - Okayama University Hospital, Okayama
  - Mie University Hospital, Tsu
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No